CLINICAL TRIAL: NCT00251628
Title: Home Care Management of Pediatric Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Kimberly A. Sutters, Kimberly A. Sutters, RN, PhD, University of California, San Francisco
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHR #H7097-14918-13; R01NR004826 (NIH)
Record Dates: First submitted 2005-11-08; First posted 2005-11-10 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Tonsillectomy
Keywords: Tonsils; Tonsillectomy
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Active Comparator)
  Interventions: Other: Standard Care; Other: As needed dosing
- Group B (Active Comparator)
  Interventions: Other: Standard Care; Other: ATC Dosing
- Group C (Experimental)
  Interventions: Other: ATC Dosing; Other: Structured Pain Management Program

INTERVENTIONS:
Other: Standard Care — standard care
  Arms: Group A; Group B
Other: ATC Dosing — ATC dosing of a weight-appropriate dose of a nonopioid/opioid combination analgesic, every 4 hours around-the-clock for the first 3 days following surgery
  Arms: Group B; Group C
Other: Structured Pain Management Program — The structured pain management program consisted of a nurse coaching intervention which included an evaluation of the child's current condition, review of the pain intensity scores, verification that the child was taking the pain medication, re-education regarding the rationale for ATC dosing, review of strategies to facilitate medication administration, and re-education about potential side effects associated with analgesic administration.
  Arms: Group C
Other: As needed dosing — "As needed" analgesic dosing with a weight-appropriate dose of a nonopioid/opioid combination analgesic, every 4 hours as needed for pain.
  Arms: Group A

SUMMARY:
The purpose of this study is to determine whether around-the-clock dosing of pain medication, with or without nurse coaching, increases the effectiveness of pain management (i.e., decreased pain intensity scores with and without swallowing, increased use of pain medication, improved sleep, increased oral intake of fluids, decreased negative behaviors, and the same degree of side effects), over time, compared to standard care with "as needed" dosing.

DETAILED DESCRIPTION:
The undertreatment of postoperative pain in children remains a critical problem. Only recently have clinical trials begun to evaluate the efficacy of pharmacologic interventions in the management of postoperative pain beyond the immediate postoperative recovery period and after discharge home following tonsillectomy. Given the fact that approximately 50% of pediatric surgeries are done on an outpatient basis, this study has the potential to improve the home pain management of thousands of children. This study is one of the first to evaluate in a systematic fashion the use of an around-the-clock dosing of a weight appropriate dose of a nonopioid/opioid combination analgesic compared to as needed dosing. Because the study will evaluate the effectiveness of both a behavioral intervention and two different pharmacologic interventions, it will provide important information that should have a direct clinical application in the management of children's pain.

The consent form is written according to the standards outlined by the Committee on Human Research, including: 1) an explanation of the purposes of the research and the expected duration of the subject's participation; 2) a description of the procedures to be followed; 3) a description of any foreseeable risks or benefits to the subject, and any alternative courses of treatment; 4) a statement describing the extent to which confidentiality of records will be maintained; 5) a statement whether compensation will be provided and medical treatment made available if injury occurs; 6) the name and number of the Chair of the Committee on Human Research; 7) a statement that participation is voluntary, and that the subject may discontinue participation at any time; and 8) a statement indicating that the subject has received a copy of the consent document and related materials. A separate form is signed to authorize access to their health care information.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient tonsillectomy, with or without other minor procedures (e.g., ear tube placement); parental consent; child assent (age-appropriate); ability of the child to speak English; ability of the parents to read, write, and speak English; and, access to a telephone.

Exclusion Criteria:

* History of severe obstructive sleep apnea (causing the child to stop breathing repeatedly during sleep); known problems with vision, hearing, control and coordination of movement, or thinking ability.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 211 (Actual)
Dates: Start 2000-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Determine the effectiveness of pain management "over time", compared to standard care with "as needed" dosing. | Morning and evening for 3 days following surgery

SECONDARY OUTCOMES:
Pain intensity | Morning and evening for 3 days following surgery
Severity of opioid-related adverse effects (i.e., nausea, vomiting, constipation, daytime sedation, lightheadedness or feeling dizzy, and nightmares) | Every evening for 3 days following surgery
Volume and number of times pain medication administered | with each dose for 3 days following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly A Sutters, RN, PhD, Principal Investigator — Children's Hospital Central California
Locations (1):
- Children's Hospital Central California, Madera, California, United States

REFERENCES:
- [Background] Sutters KA, Miaskowski C, Holdridge-Zeuner D, Waite S, Paul SM, Savedra MC, Lanier B. A randomized clinical trial of the effectiveness of a scheduled oral analgesic dosing regimen for the management of postoperative pain in children following tonsillectomy. Pain. 2004 Jul;110(1-2):49-55. doi: 10.1016/j.pain.2004.03.008. PMID 15275751
- [Background] Sutters KA, Miaskowski C, Holdridge-Zeuner D, Waite S, Paul SM, Savedra MC, Lanier B. Time-contingent dosing of an opioid analgesic after tonsillectomy does not increase moderate-to-severe side effects in children. Pain Manag Nurs. 2005 Jun;6(2):49-57. doi: 10.1016/j.pmn.2005.01.001. PMID 15970918
- [Background] Sutters KA, Savedra MC, Miaskowski C, Holdridge-Zeuner D, Waite S, Paul SM, Lanier B. Children's expectations of pain, perceptions of analgesic efficacy, and experiences with nonpharmacologic pain management strategies at home following tonsillectomy. J Spec Pediatr Nurs. 2007 Jul;12(3):139-48. doi: 10.1111/j.1744-6155.2007.00107.x. PMID 17594294
- [Background] Sutters KA, Holdridge-Zeuner D, Waite S, Paul SM, Savedra MC, Lanier B, Mahoney K, Miaskowski C. A descriptive feasibility study to evaluate scheduled oral analgesic dosing at home for the management of postoperative pain in preschool children following tonsillectomy. Pain Med. 2012 Mar;13(3):472-83. doi: 10.1111/j.1526-4637.2011.01324.x. Epub 2012 Feb 7. PMID 22313591
- [Result] Sutters KA, Miaskowski C, Holdridge-Zeuner D, Waite S, Paul SM, Savedra MC, Lanier B, Mahoney K. A randomized clinical trial of the efficacy of scheduled dosing of acetaminophen and hydrocodone for the management of postoperative pain in children after tonsillectomy. Clin J Pain. 2010 Feb;26(2):95-103. doi: 10.1097/AJP.0b013e3181b85f98. PMID 20090434
- [Result] Sutters KA, Savedra MC, Miaskowski C. The pediatric PRO-SELF(c): pain control program: an effective educational program for parents caring for children at home following tonsillectomy. J Spec Pediatr Nurs. 2011 Oct;16(4):280-94. doi: 10.1111/j.1744-6155.2011.00299.x. Epub 2011 Aug 12. PMID 21951354